CLINICAL TRIAL: NCT06602622
Title: Change in Body Weight and BMI in PWH Virologically Suppressed Who Maintain a Second-generation INSTI Regimen Compared to Those Who Switch to DOR/3TC/TDF At 48 Weeks
Brief Title: Change in Body Weight and BMI in PWH with DOR/3TC/TDF Compared with INSTI
Acronym: TLATOANI
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Principal Investigator, José Antonio Mata Marín, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2024-3502-205
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: HIV; HIV Associate Weight Loss; HIV-1 Infection; Integrase Inhibitors, HIV; HIV PROTEASE INHIB; Weight Change; Weight Loss
Keywords: HIV; Integrase inhibitors; doravirine; Body Mass Index; Body Weight Changes
MeSH Terms: conditions — Body Weight Changes; Weight Loss | interventions — Integrase Inhibitors; doravirine; Tenofovir; Lamivudine

STUDY DESIGN:
Intervention Model Description: Open label, randomized, clinical trial. Individuals who meet the inclusion criteria will be randomized to maintain their integrase inhibitor regimen (BIC/TAF/FTC, DTG/ABC/3TC or DTG+TDF/FTC) or to DOR/TDF/3TC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Integrase inhibitors (Active Comparator): Second generation integrase inhibitor: 1) Bictegravir 50 mg/ alafenamide tenofovir 25 mg/ emtricitabine 200 mg (BIC/TAF/FTC) 2) Dolutegravir 50 mg/ abacavir 600 mg/ lamivudine 300 mg (DTG/ABC/3TC) or ) dolutegravir 50 mg+ disoproxil fumarate tenofovir/ emtricitabine 300mg/ 200 mg (DTG+TDF/FTC) Each will be prescribed one tablet every day during 48 weeks
  Interventions: Drug: Integrase inhibitor
- DOR/TDF/3TC (Experimental): Individuals who meet the selection criteria will be randomized to maintain their same regimen with second-generation integrase inhibitors or switch to Doravirine/Tenofovir Disoproxil Fumarate/Emtricitabine 100/300/300 mg (DOR/TDF/3TC) It will be prescribed one tablet every day during 48 weeks
  Interventions: Drug: Doravirine + tenofovir DF + lamivudine

INTERVENTIONS:
Drug: Integrase inhibitor — Second generation integrase inhibitor 1) Bictegravir 50 mg/ alafenamide tenofovir 25 mg/ emtricitabine 200 mg (BIC/TAF/FTC); 2) Dolutegravir 50 mg/ abacavir 600 mg/ lamivudine 300 mg (DTG/ABC/3TC); 3) DTG 50mg+TDF 300mg/FTC 200mg (DTG+TDF/FTC) Each will be prescribed one tablet every day during 48 weeks
  Arms: Integrase inhibitors
Drug: Doravirine + tenofovir DF + lamivudine — Individuals who meet the selection criteria will be randomized to maintain their same regimen with second-generation integrase inhibitors or switch to DOR/TDF/3TC 100/ 300/300 mg It will be prescribed one tablet every day during 48 weeks
  Arms: DOR/TDF/3TC

SUMMARY:
Patients who developed metabolic syndrome after initiation of HIV treatment or with antiretroviral therapy (ART) for at least 36 months, treated with second generation integrase inhibitors (BIC/TAF/FTC, DTG/ABC/3Tc or DTG+TDF/FTC) who have gained at least 10% of their total body weight after starting ART, with a body mass index ≥25 kg/m2 and body fat greater than 20% will be eligible to participate in this clinical trial. If they decide to participate, they will sign an informed consent. After this, a mobile application will randomly decide whether the participant will continue with their ART regimen or switch to another ART (listed in the guidelines as one of the main lines of treatment) containing doravirine/lamivudine/disoproxil fumarate tenofovir. Medical visits will be at 1 month, 3 months, 6 months, 9 months, and 12 months after get in to this protocol, with laboratory studies that evaluate fats, blood sugar, liver function, kidney function, and test for HIV control; in addition, each visit will be given self-fillable scales to evaluate neuropsychiatric disorders such as depression, anxiety, insomnia, satisfaction with treatment or symptoms associated with it.The aim of the study is to observe whether there is weight loss with the change in HIV treatment.

DETAILED DESCRIPTION:
Open-label, randomized clinical trial, conducted at the infectious disease hospital, La Raza National Medical Center, Mexico City, from July 2024 to November 2025.

The aim of the study is to determine the percentage change in body weight and BMI in virologically suppressed PWH maintaining a second-generation INSTI (BIC/TAF/FTC, DTG/ABC/3TC or DTG+TDF/FTC) regimen compared with those switching to DOR/3TC/TDF at 48 weeks post-switch.

PWH who are on a second-generation INSTI regimen who are virologically suppressed (HIV-1 RNA minor to 50 copies/mL) and have gained ≥10% of their body weight compared to their weight before starting ART, BMI ≥25 kg/m2, and body fat greater than 20% will be identified, and invited to participate.

A medical interview will be conducted to assess clinical characteristics, comorbidities of the study subject, new drugs, changes in doses or suspensions, as well as plans by their other physicians for changes in the same, diet, frequency and intensity of exercise. Once the preliminary information has been obtained, it will be established whether the patient is a candidate to take part in the study and will be invited to participate voluntarily. The project and the probable results, benefits and risks of participating will be explained in detail and in detail; If they agree to participate, informed consent will be obtained from the principal investigator or associate researchers during the medical visit where weight gain and BMI are identified, for authorization to take clinical exams, anthropometric measurements (these will be carried out by the principal investigator or associates). A response will be obtained during the same medical visit with free decision to continue or withdraw from the study at the time deemed appropriate during the study period without this affecting your medical care at the HIV clinic. (Annex 1) Patients who accept will be asked again for HIV-1 RNA, CD4+, complete blood count, lipid profile, complete liver enzymes, cystatin C and urinary electrolytes within 45 days prior to randomization, and if they meet the inclusion criteria, through simple randomization and with the randomizer for clinical trial application, the principal investigator will randomize them into the group of maintaining the previous regimen with second-generation INSTI or changing the regimen to DOR/3TC/TDF, and in order to maintain privacy, a folio number will be assigned at the time of recruitment.

Weight measurements will be taken with a FitScan segmental body composition monitor BC-545F scale, height in centimeters, body mass index (BMI) with the formula weight (kg)/height (m2), body composition (fat in %, water in %, muscle in kg, bone in kg) with a FitScan segmental body composition monitor BC-545F equipment, waist and hip measurements with a measuring tape in cm.

Laboratory studies will include complete blood count, complete blood chemistry with glucose, creatinine, complete lipid profile, and liver function tests after randomization at 4 weeks, 12 weeks, 24 weeks, and 48 weeks post-switch. CD4+, HIV-1 RNA, Cystatin C, and urinary electrolytes will be determined prior to randomization, at 6 months, and 12 months after entering the study. Comparisons will be made between measurements taken prior to entering the study, at 24 and 48 weeks after entering the study.

In case of elevated AST and/or ALT &amp;gt;90 IU/L, serologies will be requested to rule out HBV and HCV.

The PSQI, ISI, HADS-A, and HADS-D questionnaires will be used to assess anxiety, depression, and sleep quality; in addition, the HIVTSQ questionnaire will be used to assess treatment satisfaction at weeks 4, 12, 24, and 48 weeks after randomization, and HIV Symptoms Distress Module (HIV-SDM).

The change in weight and BMI at 48 weeks will be defined as the difference between the weight and BMI prior to randomization compared to the results at 48 weeks, weight will be expressed in kg, percentages and BMI in kg/m2.

The sampling was simple random, participation in the study was offered to all Mexican patients living with HIV who have gained ≥10% of body weight and BMI ≥25% from a regimen with second-generation integrase inhibitor (BIC/TAF/FTC or DTG/ABC/3TC).

Sample size per group: 54 participants per group. Calculated based on the expected change after switching from INSTI to a regimen with DOR/TDF/3TC, with estimated losses of 20%, 108 participants in total.

Kolmogorov-Smirnoff test will be used to identify distribution of data and to express central tendency measures (medians with interquartile ranges) and percentages accordingly. Data will be compared using the Mann-Whitney U test. Qualitative data will be analyzed using the x2 or Fisher´s exact test, as appropriate. Subsequently, data will be analyzed by groups at 12, 24, 36, and 48 weeks using the Wilcoxon test. A P value ≤0.05 with a 95% confidence interval will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Virologically suppressed for at least 48 weeks prior to study entry
2. Coming from a regimen containing Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/FTC/TAF), Dolutegravir/Lamivudine/Abacavir (DTG/3TC/ABC), or, Dolutegravir/Tenofovir Disoproxil Fumarate/Emtricitabine (DTG+TDF/FTC) with no known failures to integrase inhibitors for al least 48 weeks.
3. BMI ≥25 kg/m2 at screening and
4. Unintentional weight gain of >10% from baseline (prior to INSTI initiation) within 1-3 years of starting INSTI ART, with no other apparent medical reason to explain the weight gain (concomitant medication use, Cushing's disease, recent prolonged hospitalization, etc.), in the opinion of the site investigator.
5. Body fat percentage >20%
6. No indication or plans to add or change medications associated with significant weight change during the study period.
7. Participants currently receiving antipsychotics, antidepressants, anticonvulsants/mood stabilizers, and thyroid replacement hormones without dose modifications for at least 12 weeks prior to randomization
8. Participants currently receiving antidiabetics known to cause weight loss and without dose modifications for at least 24 weeks prior to randomization (GLP-1 receptor agonists, SGLT-2 inhibitors, insulin, metformin).
9. Agree to adhere to assigned ART during the study period
10. HIV-1 RNA screening <50 copies/mL performed within 45 days prior to study entry.
11. GFR by CDK-EPI ≥60 mL/min
12. Alanine aminotransferase (ALT) and asparatate aminotransferase (AST) < 90 IU/L
13. Thyroid profile (TSH, free T3 and free T4) prior to entering the study
14. Serum and urinary electrolytes, cystatin C, prior to entering the study

Exclusion Criteria:

1. Loss of social security
2. Allergy to any of the components of ART, previously unknown.
3. Withdrawal of informed consent
4. Acquiring HBV and/or HCV infection during follow-up.
5. HIV-1 RNA >200 copies/mL in 2 consecutive determinations after having achieved virological suppression.
6. Early initiation or discontinuation of any of the following drugs after entering the study: antipsychotics (clozapine, olanzapine, risperidone); antidepressants (tricyclic antidepressants, selective serotonin reuptake inhibitors) monoamine oxidase inhibitors, associated with weight gain; anticonvulsants/mood stabilizers (lithium, valproic acid) or associated with weight loss (topiramate); thyroid replacement hormones;
7. Change in dose or discontinuation of antidiabetic drugs that cause weight loss (GLP-1 receptor agonists, SGLT-2 inhibitors, insulin, metformin), after entering the study.
8. Planning to undergo or having undergone bariatric surgery.
9. Initiating significant dietary changes, advised by a nutritionist according to what was reported by the participant
10. Initiating or increasing physical exercise or enrolling in a structured weight loss regimen: <250 minutes/week of moderate to intense activity

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-11-14 (Estimated); Study Completion 2025-11-14 (Estimated)

PRIMARY OUTCOMES:
Change in body weight and BMI | 48 weeks
  To determine the percentage change in body weight and BMI in virologically suppressed PLHIV maintaining a second-generation INSTI regimen compared with those switching to DOR/3TC/TDF at 48 weeks post-switch. This will be measured with with the same scale at baseline, 1 month, 3 months, 6 months, 9 months and 12 months.

SECONDARY OUTCOMES:
Adverse events | 48 weeks
  Evaluate the number and degree of adverse events in each group of ART at baseline, 1 month, 3 months, 6 months, 9 months and 12 months post-recruitment
Evaluate neuropsychiatric disorders | 48 weeks
  Assess sleep quality using the Insomnia Severity Score (ISI) baseline and at 48 weeks Assess anxiety and depression using the Hospital Anxiety and Depression Scales (HADS-A and HADS-D) baseline and at 48 weeks Assess the presence and degree of depression using the Patient Health Questionnaire-9 (PHQ-9) baseline and at 48 weeks. This will be measured at baseline, 1 month, 3 months, 6 months, 9 months and 12 months.
Changes in lipid profile | 48 weeks
  Analyze changes in total cholesterol, hdl cholesterol and triglycerides at baseline and 48 weeks after switch. This will be evaluated at baseline, 1 month, 3 months, 6 months, 9 months and 12 months.
Analyze changes in body composition | 48 weeks
  Fat in percentage, muscle in kilograms, water in percentage and bone in kilograms. This will be evaluated with same bioimpedance equipment at baseline, 1 month, 3 months, 6 months, 9 months and 12 months.
Cardiovascular risk | 48 weeks
  Determine cardiovascular risk using Framingham scale and Atherosclerotic Cardiovascular Disease. (ASCVD) at baseline an 48 weeks. This will be evaluated at baseline, 6 months, and 12 months.
Kidney function | 48 weeks
  Analyze changes in renal function using creatinine, cystatin C, and urinary electrolytes at baselina and 48 weeks. This will be evaluated at baseline, 6 months, and 12 months.

OTHER OUTCOMES:
HIVSDM scale symptom distress scale | 48 weeks
  Symptom distress an instrument to identify perceived individual symptoms reported by HIV infected patients. The construct distress, in an HIV population, is characterized by phenomena such as fatigue/low energy, fevers, dizziness, tingling/hand/foot pain, memory loss, nausea/vomiting, diarrhea, depression, anxiety, sleep problems, skin problems, cough/shortness of breath, headache, appetite loss, bloating/gas, muscle/joint pain, sexual problems, weight gain weight loss, and hair loss. This will be measured at baseline, 1 month, 3 months, 6 months, 9 months and 12 months.
HIV Treatment Satisfaction Questionnaire (HIVTSQ) | 48 weeks
  The HIV treatment Satisfaction Questionnaire is a Patient-reported questionnaire that assesses treatment satisfaction, specific to patients with HIV-1. Is a10-item self-answered where they are asked to respond to each of 10 questions, by circling a number (0-6), this will be measured at baseline, 1 month, 3, 6, 9 and 12 months after switch.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de infectología, Centro Médico Nacional La Raza, Mexico City, Azcapotzalco, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be shared if necessary, as it contains personal and sensitive information about participants.

REFERENCES:
- [Background] O'Halloran JA, Sahrmann J, Parra-Rodriguez L, Vo DT, Butler AM, Olsen MA, Powderly WG. Integrase Strand Transfer Inhibitors Are Associated With Incident Diabetes Mellitus in People With Human Immunodeficiency Virus. Clin Infect Dis. 2022 Dec 19;75(12):2060-2065. doi: 10.1093/cid/ciac355. PMID 35521785
- [Background] Orkin C, Squires KE, Molina JM, Sax PE, Wong WW, Sussmann O, Kaplan R, Lupinacci L, Rodgers A, Xu X, Lin G, Kumar S, Sklar P, Nguyen BY, Hanna GJ, Hwang C, Martin EA; DRIVE-AHEAD Study Group. Doravirine/Lamivudine/Tenofovir Disoproxil Fumarate is Non-inferior to Efavirenz/Emtricitabine/Tenofovir Disoproxil Fumarate in Treatment-naive Adults With Human Immunodeficiency Virus-1 Infection: Week 48 Results of the DRIVE-AHEAD Trial. Clin Infect Dis. 2019 Feb 1;68(4):535-544. doi: 10.1093/cid/ciy540. PMID 30184165
- [Background] Calza L, Giglia M, Colangeli V, Bon I, Vitale S, Viale P. Improvement in insulin sensitivity after switching from an integrase inhibitor-based regimen to doravirine/tenofovir disoproxil fumarate/lamivudine in people with significant weight gain. HIV Med. 2024 Aug;25(8):919-926. doi: 10.1111/hiv.13644. Epub 2024 Apr 3. PMID 38570897
- [Background] Orkin C, Elion R, Thompson M, Rockstroh JK, Alvarez Bognar F, Xu ZJ, Hwang C, Sklar P, Martin EA. Changes in weight and BMI with first-line doravirine-based therapy. AIDS. 2021 Jan 1;35(1):91-99. doi: 10.1097/QAD.0000000000002725. PMID 33048879
- [Background] Molina JM, Squires K, Sax PE, Cahn P, Lombaard J, DeJesus E, Lai MT, Xu X, Rodgers A, Lupinacci L, Kumar S, Sklar P, Nguyen BY, Hanna GJ, Hwang C; DRIVE-FORWARD Study Group. Doravirine versus ritonavir-boosted darunavir in antiretroviral-naive adults with HIV-1 (DRIVE-FORWARD): 48-week results of a randomised, double-blind, phase 3, non-inferiority trial. Lancet HIV. 2018 May;5(5):e211-e220. doi: 10.1016/S2352-3018(18)30021-3. Epub 2018 Mar 25. PMID 29592840
- [Background] Bares SH, Wu X, Tassiopoulos K, Lake JE, Koletar SL, Kalayjian R, Erlandson KM. Weight Gain After Antiretroviral Therapy Initiation and Subsequent Risk of Metabolic and Cardiovascular Disease. Clin Infect Dis. 2024 Feb 17;78(2):395-401. doi: 10.1093/cid/ciad545. PMID 37698083
- [Background] Sokhela S, Venter WDF, Bosch B, Woods J, McCann K, Akpomiemie G, Chandiwana N, Mashabane N, Tembo A, Simmons B, Lalla-Edward S, Siedner MJ, Sinxadi P, Hermans L, Fairlie L, Vos A, Abrams E, Manne-Goehler JM, Moorhouse M, Clayden P, Norris S, Qavi A, Chersich M, Masenya M, Arulappan N, Hill A. Final 192-Week Efficacy and Safety Results of the ADVANCE Trial, Comparing 3 First-line Antiretroviral Regimens. Open Forum Infect Dis. 2024 Jan 24;11(3):ofae007. doi: 10.1093/ofid/ofae007. eCollection 2024 Mar. PMID 38529213
- [Background] Gadde KM, Martin CK, Berthoud HR, Heymsfield SB. Obesity: Pathophysiology and Management. J Am Coll Cardiol. 2018 Jan 2;71(1):69-84. doi: 10.1016/j.jacc.2017.11.011. PMID 29301630
- [Background] Eckard AR, McComsey GA. Weight gain and integrase inhibitors. Curr Opin Infect Dis. 2020 Feb;33(1):10-19. doi: 10.1097/QCO.0000000000000616. PMID 31789693
- [Background] Hogg RS, Eyawo O, Collins AB, Zhang W, Jabbari S, Hull MW, Lima VD, Ahmed T, Kendall CE, Althoff KN, Justice AC, Barrios R, Shoveller J, Montaner JSG; Comparative Outcomes And Service Utilization Trends (COAST) study. Health-adjusted life expectancy in HIV-positive and HIV-negative men and women in British Columbia, Canada: a population-based observational cohort study. Lancet HIV. 2017 Jun;4(6):e270-e276. doi: 10.1016/S2352-3018(17)30029-2. Epub 2017 Mar 3. PMID 28262574
- [Background] Marcus JL, Leyden WA, Alexeeff SE, Anderson AN, Hechter RC, Hu H, Lam JO, Towner WJ, Yuan Q, Horberg MA, Silverberg MJ. Comparison of Overall and Comorbidity-Free Life Expectancy Between Insured Adults With and Without HIV Infection, 2000-2016. JAMA Netw Open. 2020 Jun 1;3(6):e207954. doi: 10.1001/jamanetworkopen.2020.7954. PMID 32539152